CLINICAL TRIAL: NCT04897776
Title: Thalamic Stimulation to Prevent Impaired Consciousness in Epilepsy
Brief Title: Stimulation of the Thalamus for Arousal Restoral in Temporal Lobe Epilepsy
Acronym: START
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Mayo Clinic (Other); Dartmouth-Hitchcock Medical Center (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Hal Blumenfeld, MD, PhD, Professor of Neuroscience and of Neurosurgery, Yale University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2000030289; 1UG3NS112826-01 (NIH)
Record Dates: First submitted 2021-05-11; First posted 2021-05-24 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-11

CONDITIONS: Epilepsy, Temporal Lobe
Keywords: Thalamic Stimulation; Hippocampal Stimulation; Awareness; Ictal Awareness; Post-ictal Awareness; Consciousness; Temporal Lobe Epilepsy; Epilepsy; Quality of Life; Cognition; Neurostimulation; Deep Brain Stimulation; Responsive Neurostimulation; Intralaminar Thalamus; Thalamic Central Lateral Nucleus; Device; Behavioral Assessment
MeSH Terms: conditions — Epilepsy, Temporal Lobe; Epilepsy

STUDY DESIGN:
Intervention Model Description: After controlling for implant effects and hippocampal stimulation, there will be a period of blinding for thalamic stimulation. Physician and patient will not know which seizures during this period receive stimulation or sham stimulation. The primary outcome measure will be comparing behavioral awareness scores during this period, sham stimulation compared to therapeutic stimulation.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Therapeutic Thalamic Stimulation (Experimental): Four months post implant, the neurostimulator device will provide patients with hippocampal stimulation for all seizures. For seizures longer than five seconds, thalamic stimulation will be administered at a therapeutic level established based on the physician's evaluation and patient specific parameters established at a previous visit. This will occur in half of the seizures the patient experiences and will be randomly assigned during this phase of the study.
  If no benefit is experienced during this phase of the study, patients may participate in an optional randomized CL stimulation phase for an additional four months.
  Interventions: Device: Central Thalamic Stimulation; Device: Hippocampal Stimulation
- Non-Therapeutic Thalamic Stimulation (Sham Comparator): Four months post implant, the neurostimulator device will provide patients with hippocampal stimulation for all seizures. For seizures longer than five seconds, thalamic stimulation will be administered at below therapeutic threshold to control for implant and placebo effects. This will occur in half of the seizures the patient experiences and will be randomly assigned during this phase of the study.
  If no benefit is experienced during this phase of the study, patients may participate in an optional randomized CL stimulation phase for an additional four months.
  Interventions: Device: Hippocampal Stimulation

INTERVENTIONS:
Device: Central Thalamic Stimulation — Stimulation of the bilateral thalamic CL is a promising approach in human patients to improve conscious arousal. To restore conscious arousal by stimulation of the thalamic intralaminar CL it is necessary to provide bilateral stimulation, placing one lead in each thalamus. Bilateral thalamic CL stimulation was shown previously to improve human conscious arousal and is based on existing research in patients with disorders of consciousness.
  Arms: Therapeutic Thalamic Stimulation
Device: Hippocampal Stimulation — The hippocampus has been a target for brain stimulation for seizure reduction in epilepsy. While the efficacy of HC stimulation varies considerably among different studies, the surgical procedure and therapeutic electrical stimulation are well tolerated by patients, with few peri-operative complications being reported, and histopathologic analysis not revealing a difference between stimulated and non-stimulated hippocampal tissue (Han et al. 2014)

SUMMARY:
The goal is to provide a novel therapeutic option for temporal lobe epilepsy patients when focal impaired awareness seizures cannot be stopped by medications, surgical or laser ablation, or by neurostimulation. The goal is restore consciousness when seizures cannot be stopped. If successful, addition of bilateral thalamic stimulation to existing responsive neurostimulation to rescue consciousness would greatly alter clinical practice and patient outcomes.

Importantly, previous approaches aim to stop seizures, whereas this study aims to use thalamic stimulation to improve a major negative consequence when seizures cannot be stopped. The potential impact extends beyond temporal lobe epilepsy to other seizure types, and may also extend more broadly to inform treatment of other brain disorders associated with impaired consciousness and cognition.

DETAILED DESCRIPTION:
Impaired consciousness during seizures has a major negative impact on quality of life for people with epilepsy. Consequences include risk of motor vehicle accidents, drowning, poor work and school performance, and social stigmatization. Impaired ictal/postictal arousal may also compromise breathing leading to sudden unexpected death in epilepsy. Although the primary goal of epilepsy care is to stop seizures, restoring conscious awareness in patients whose seizures cannot be stopped (by medications, surgery or deep brain stimulation) could significantly improve outcome. Disorders of consciousness other than epilepsy have long been known to arise from dysfunction of subcortical-cortical arousal circuits. Deep brain stimulation (DBS) of the thalamic intralaminar central lateral nuclei (CL) is a promising approach to restore conscious arousal currently being trialed for chronic disorders of consciousness. Recent neuroimaging and EEG studies have shown that transient impaired consciousness in temporal lobe epilepsy (TLE) seizures also depends on subcortical-cortical arousal including thalamic CL. Translational studies from this research group further demonstrate depressed CL function in limbic seizures, and most importantly that thalamic CL stimulation has the potential to restore physiological and behavioral arousal in the ictal and postictal periods. DBS treatment of epilepsy has advanced rapidly with FDA approval of responsive neurostimulation (RNS, NeuroPace) and thalamic anterior nucleus stimulation (Medtronic). Investigational devices such as the Medtronic Summit RC+S provide a unique opportunity for responsive stimulation of up to four separate brain regions, enabling conventional sites such as hippocampus (HC) to be combined with innovative targets such as thalamic CL. Meanwhile, collaborators Mayo Clinic have developed the Epilepsy Personal Assistant Device (EPAD), a custom application running on a hand-held device with bi-directional communication with the RC+S. The EPAD will enable cloud-based data storage, seizure diaries, and automatic behavioral tests. Therefore, the goal is to develop and pilot test the feasibility and safety of bilateral thalamic CL stimulation using RC+S to restore conscious arousal in TLE seizures which are not stopped by conventional responsive neurostimulation, offering hope to greatly improve quality of life in these patients.

ELIGIBILITY:
Inclusion Criteria:

1. All patients will have evidence of mesial temporal seizures based on either

   1. Intracranial EEG monitoring with mesial temporal lobe onset
   2. or scalp EEG evidence of temporal lobe seizures and other evidence of mesial temporal lobe epilepsy.
2. Subject's seizure focus, based upon clinical history, semiology, electroencephalographic (EEG) findings, and/or neuroimaging, shall demonstrate bilateral or unilateral mesial temporal lobe epilepsy, and subject shall not be good candidate for surgical resection.
3. Focal epilepsy with disabling seizure counts mean of ≥ 2 per month. Disabling seizures are those with significant negative impact on the patient's life, involving impaired conscious awareness. Seizures counts will be based on patient's self-report. Note that patient's typically have more disabling seizures than they are able to self-report, and may also have additional non-disabling seizures in addition to the disabling seizures required for enrolment.

   i. Mean seizure count ≥ 2 per month is established initially for the preceding 6 months at time of Enrollment, using seizures reported by the patient and/or caregiver. Seizures during EMU admissions are not included.
4. Drug resistance to at least two antiseizure medications (ASM) with adequate dose and duration.
5. Subject is willing to remain on stable ASM from the Baseline phase through the end of the Randomized CL Stimulation phase. Stable is defined as same medications, but dose adjustments are allowed within accepted therapeutic ranges. Also, short-term benzodiazepines allowed for acute seizure worsening as in prior studies.
6. Apart from epilepsy, subject must be medically and neurologically stable and must have no other medical condition in the opinion of the treating physician that would preclude the patient from participation. This could include conditions like severe ischemic cardiac disease, progressive dementia or other disorders that could affect surgical eligibility or compliance.
7. The local treating epilepsy center has recommended the patient for brain stimulation therapy on clinical grounds and without reference to this protocol.
8. Age 18 to 75 years, inclusive, at time of consent.
9. Ability and willingness to provide informed consent and participate in the study protocol.
10. Subject can interpret and to respond, in accordance with the study protocol, to the advisory indicators provided by the device. This includes the ability to recharge the device.
11. Subject has seizures that are distinct, stereotypical events that can be reliably counted by the patient or caregiver.
12. Subject can reasonably be expected to maintain a seizure diary alone or with the assistance of a competent individual.
13. Subject can complete regular office visits and telephone appointments in accordance with the study protocol requirements.
14. A female subject must have a negative pregnancy test and if sexually active, must be using a reliable form of birth control for the duration of the trial, be surgically sterile, or be at least two years post-menopausal.
15. Subject has been informed of his or her eligibility for resective surgery as a potential alternative to the study, if such surgery is a reasonable option.
16. Subject speaks and reads English.
17. Subject's anatomy will permit implantation of the Medtronic Investigational Summit RC+S generator within 20 mm of the skin surface.
18. Subject is capable of completing the proposed neuropsychology evaluation and will score no lower than 2 standard deviations below average on the Wechsler Adult Intelligence Scale.

Exclusion Criteria:

1. Subject has a contraindication to magnetic resonance imaging.
2. Subject has a significant substance abuse history (alcohol, prescription, or illicit medications) within the preceding two years with evidence of impact on daily function.
3. Subject participated in another drug or device trial within the preceding 30 days.
4. Demonstrates that they fulfill criteria on any of the three subscale of the SCID-5-PD for borderline, antisocial, or narcissistic personality disorders and these criteria are then corroborated by psychiatric interview, and that this would significantly affect participation in the study.
5. Suicide attempt in the past year.
6. Arrest for assault or possession of drugs or weapons with intent to sell/distribute in the past year.
7. Subject is implanted with pacemaker, implantable cardiac defibrillator, cardiac management product, or a medical device that interferes with the RC+S device. This includes, but is not limited to, direct brain neurostimulators, spinal cord stimulators, vagus nerve stimulators (VNS), and cochlear implants. Patients with a vagus nerve stimulator implanted but turned off through the duration of the study may be enrolled, provided their clinical status has been stable for at least one month with VNS turned off. Alternatively, patients with a VNS may have the previously disabled VNS removed at time of surgery to implant the Medtronic RC+S.
8. Subject has confirmed active diagnosis of psychogenic or non-epileptic seizures.
9. Subject has confirmed diagnosis of primary generalized seizures.
10. Subject has experienced unprovoked status epilepticus in the preceding year.
11. Subject has had therapeutic surgery to treat epilepsy that may interfere with electrode placement.
12. Subject has progressive neurological disorder or medical condition that would prevent the participant to fully participate in the clinical trial.
13. Subject has severe chronic pulmonary disease or cardiac disease, local, systemic acute or chronic infectious illness.
14. Subject is on anticoagulants and is unable to discontinue them peri-surgically, as required by the neurosurgeon or Investigator.
15. Subject has significant platelet dysfunction from medical conditions or medications (including, particularly, aspirin or sodium valproate). If platelet dysfunction is suspected, subject can be enrolled only if a hematologist, the Investigator, and the neurosurgeon judge it to be advisable.
16. Subject is ineligible for cranial surgery.
17. Subject scores equal to or below a full-scale intelligence quotient (FSIQ) of 70, as measured by the Wechsler Adult Intelligence Scale.
18. Pregnancy.
19. Any condition or finding that in the judgement of the site PI significantly increases risk or significantly reduces the likelihood of benefit from participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-10-31 (Actual); Primary Completion 2025-06-16 (Actual); Study Completion 2025-07-15 (Actual)

PRIMARY OUTCOMES:
Change in Conscious Awareness | Up to 45 months
  Evaluate levels of conscious awareness during and following seizures, based on a behavioral responsiveness scale. Behavioral responsiveness is delivered on a tablet device automatically when a seizure is identified by the neurostimulator device. Automatic Responsiveness Testing in Epilepsy has a score range of 0 to 18, where 0 is not consciousness and/or unable to interact appropriately to commands and 18 is conscious, aware, and able to interact appropriately to commands. This is measured at scheduled in weekly intervals prior to implant and continuously over the 45 months of participation that occur post-implant.

SECONDARY OUTCOMES:
Change in Seizure Severity | Up to 45 months
  Evaluate changes seizure severity with the Liverpool Seizure Severity Questionnaire. Questionnaires will be given to patients to complete during in-person visits to evaluate changes in reported seizure frequency, which will also be compared to the objective seizure count from the Medtronic Summit RC+S device post-implant. The Liverpool Seizure Severity Scale 2.0 questionnaire produces a single unit-weighted scale that measures severity of the most severe seizures the patient experienced during the recall period. Score ranges are from 0 to 100, where 0 is the patient reports no seizures whereas 100 indicates frequent seizures with severe symptomology, including headaches, confusion, and delays in returning to tasks. Measured at each in-person visit from Baseline to End of Study (13 times over 45 months).
Change in Quality of Life | Up to 45 months
  Evaluate changes quality of life periodically with epilepsy-specific standardized assessment tools. Questionnaire will be given to patients to complete at in-person visits as to evaluate changes in quality of life. Quality of Life in Epilepsy Inventory is converted to a t-score range of 11 to 73, where 11 is a low quality of life with limited independence, low cognitive function, and significant seizure worry whereas a score of 73 indicates high levels of satisfaction in their health, minimal seizure worry, and high social function. Measured at each in-person visit from Baseline to End of Study (13 times over 45 months).

OTHER OUTCOMES:
Change in Seizure Frequency | Up to 45 months
  Monitor seizure frequency with use of seizure diaries prior to neurostimulator implant and continuous monitoring from the Medtronic Summit RC+S once implanted.

CONTACTS AND LOCATIONS:
Overall Officials: Hal Blumenfeld, MD, PhD, Principal Investigator — Yale University; Barbara Jobst, MD, PhD, Principal Investigator — Dartmouth-Hitchcock Medical Center; Gregory Worrell, MD, PhD, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Yale New Haven Hospital, New Haven, Connecticut
  - Mayo Clinic, Rochester, Minnesota
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Han CL, Hu W, Stead M, Zhang T, Zhang JG, Worrell GA, Meng FG. Electrical stimulation of hippocampus for the treatment of refractory temporal lobe epilepsy. Brain Res Bull. 2014 Oct;109:13-21. doi: 10.1016/j.brainresbull.2014.08.007. Epub 2014 Sep 6. PMID 25200252
- [Background] Geller EB, Skarpaas TL, Gross RE, Goodman RR, Barkley GL, Bazil CW, Berg MJ, Bergey GK, Cash SS, Cole AJ, Duckrow RB, Edwards JC, Eisenschenk S, Fessler J, Fountain NB, Goldman AM, Gwinn RP, Heck C, Herekar A, Hirsch LJ, Jobst BC, King-Stephens D, Labar DR, Leiphart JW, Marsh WR, Meador KJ, Mizrahi EM, Murro AM, Nair DR, Noe KH, Park YD, Rutecki PA, Salanova V, Sheth RD, Shields DC, Skidmore C, Smith MC, Spencer DC, Srinivasan S, Tatum W, Van Ness PC, Vossler DG, Wharen RE Jr, Worrell GA, Yoshor D, Zimmerman RS, Cicora K, Sun FT, Morrell MJ. Brain-responsive neurostimulation in patients with medically intractable mesial temporal lobe epilepsy. Epilepsia. 2017 Jun;58(6):994-1004. doi: 10.1111/epi.13740. Epub 2017 Apr 11. PMID 28398014
- [Background] Salanova V, Witt T, Worth R, Henry TR, Gross RE, Nazzaro JM, Labar D, Sperling MR, Sharan A, Sandok E, Handforth A, Stern JM, Chung S, Henderson JM, French J, Baltuch G, Rosenfeld WE, Garcia P, Barbaro NM, Fountain NB, Elias WJ, Goodman RR, Pollard JR, Troster AI, Irwin CP, Lambrecht K, Graves N, Fisher R; SANTE Study Group. Long-term efficacy and safety of thalamic stimulation for drug-resistant partial epilepsy. Neurology. 2015 Mar 10;84(10):1017-25. doi: 10.1212/WNL.0000000000001334. Epub 2015 Feb 6. PMID 25663221
- [Background] Schiff ND, Giacino JT, Kalmar K, Victor JD, Baker K, Gerber M, Fritz B, Eisenberg B, Biondi T, O'Connor J, Kobylarz EJ, Farris S, Machado A, McCagg C, Plum F, Fins JJ, Rezai AR. Behavioural improvements with thalamic stimulation after severe traumatic brain injury. Nature. 2007 Aug 2;448(7153):600-3. doi: 10.1038/nature06041. PMID 17671503
- [Background] Kremen V, Brinkmann BH, Kim I, Guragain H, Nasseri M, Magee AL, Pal Attia T, Nejedly P, Sladky V, Nelson N, Chang SY, Herron JA, Adamski T, Baldassano S, Cimbalnik J, Vasoli V, Fehrmann E, Chouinard T, Patterson EE, Litt B, Stead M, Van Gompel J, Sturges BK, Jo HJ, Crowe CM, Denison T, Worrell GA. Integrating Brain Implants With Local and Distributed Computing Devices: A Next Generation Epilepsy Management System. IEEE J Transl Eng Health Med. 2018 Sep 26;6:2500112. doi: 10.1109/JTEHM.2018.2869398. eCollection 2018. PMID 30310759
- See also: Mayo Clinic Appointment Request — https://onlineservices.mayoclinic.org/NewAppointments/
- See also: Yale University Appointment Request — https://www.yalemedicine.org/departments/epilepsy-and-seizures
- See also: Dartmouth-Hitchcock Medical Center Appointment Request — https://www.dartmouth-hitchcock.org/epilepsy/appointments-referrals